CLINICAL TRIAL: NCT04071379
Title: Comparison of Immunogenicity and Safety of DTP-HB-Hib (Bio Farma) With Pentabio® Vaccine Primed With Recombinant Hepatitis B at Birth Dose (Using Different Source of Hepatitis B), in Indonesian Infants
Brief Title: Comparison of Immunogenicity and Safety of DTP-HB-Hib (Bio Farma) With Pentabio® Vaccine Primed With Recombinant Hepatitis B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Penta BS19
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Immunogenicity; Safety

STUDY DESIGN:
Intervention Model Description: Subjects neonates: Randomized, double blind, 2 arms parallel groups, prospective intervention Study
Who Masked: Participant, Investigator
Masking Description: Randomized, double blind, 2 arms parallel group, prospective intervention study This study will do the lot to lot consistency and will be compared to registered product
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HepB + Penta batch 1 (Experimental): Recombinant Hepatitis B + DTP-HB-Hib batch 1
  Interventions: Biological: Recombinant Hepatitis B + DTP-HB-Hib
- Hep B + Pentabio (registered) (Active Comparator): Recombinant Hepatitis B + Pentabio (registered)
  Interventions: Biological: Hep B + Pentabio (registered)

INTERVENTIONS:
Biological: Recombinant Hepatitis B + DTP-HB-Hib — 1 dose of 0.5 ml Recombinant Hepatitis B + 3 dose of 0.5 ml of DTP-HB-Hib
  Other Names: Hep B + DTP-HB-Hib
  Arms: HepB + Penta batch 1
Biological: Hep B + Pentabio (registered) — 1 dose of 0.5 ml Recombinant Hepatitis B (registered) + 3 dose of 0.5 ml of Pentabio (registered)
  Other Names: Recombinant Hepatitis B (Bio Farma) + Pentabio (Bio Farma)
  Arms: Hep B + Pentabio (registered)

SUMMARY:
Comparison of Immunogenicity and Safety of DTP-HB-Hib (Bio Farma) with Pentabio® vaccine Primed with Recombinant Hepatitis B

DETAILED DESCRIPTION:
Comparison of Immunogenicity and Safety of DTP-HB-Hib (Bio Farma) with Pentabio® vaccine Primed with Recombinant Hepatitis B at Birth dose (using different source of Hepatitis B), in Indonesian Infants

ELIGIBILITY:
Inclusion Criteria:

* Healthy, full term, newborns infants.
* Infant born after 37-42 weeks of pregnancy.
* Infant weighing 2500 gram or more at birth.
* Father, mother or legally acceptable representative properly informed about the study and having signed the informed consent form.
* Parents will commit themselves to comply with the indications of the investigator and with the schedule of the trial.

Exclusion Criteria:

* Child concomitantly enrolled or scheduled to be enrolled in another trial.
* Mother with HBsAg positive.
* Evolving mild, moderate or severe illness, especially infectious diseases or fever (axillary temperature >37.5C on Day 0).
* Suspected of allergy to any component of the vaccines (e.g. formaldehyde).
* Suspected of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection.
* Newborn suspected of congenital or acquired immunodeficiency (including HIV infection).
* Received or plans to receive any treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products or long term corticotherapy (> 2 weeks)).
* Received other vaccination with the exception of BCG and poliomyelitis.
* Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives.

Ages: 0 Days to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
To evaluate protectivity of DTP-HB-Hib Vaccine (Bio Farma) with new Hepatitis B bulk | 28 days after immunization
  Percentage of infants with anti-diphtheria titer and anti-tetanus titer > 0.01 IU/ml, anti HbsAg titer > 10 mIU/ml, and anti PRP-T titer > 0.15 ug/ml 28 days after the last injection of DTP/HB/Hib with different source of Hepatitis B bulk vaccine group.

SECONDARY OUTCOMES:
Describes antibody response to diphtheria toxoid, tetanus toxoid in both group with the evaluation criteria | 28 days after immunization
  Serological response to diphtheria toxoid, tetanus toxoid: GMT, percentage of infants with titer > 0.01 IU/ml, > 0.1 IU/ml percentage of infants with increasing antibody titer > 4 times and/or percentage of infants with transition of seronegative to seropositive
Serological response to the pertussis component (agglutinins) | 28 days after immunization
  Serological response to the pertussis component (agglutinins): GMT, percentage of infants with titer > 40, > 80, > 160 and > 320 (1/dil.), percentage of infants with increasing antibody titer > 4 times
Geometric mean of anti-HbsAg | 28 days after immunization
  Geometric mean of anti-HbsAg, percentage of infants with titer > 10mIU/ml, percentage of infants with increasing antibody titer > 4 times and/ or percentage of infants with transition of seronegative to seropositive
Serological response to Hib/PRP | 28 days after immunization
  Serological response to Hib/PRP: GMT, percentage of infants with titer >1 ug /ml ; > 0.15 ug /ml percentage of infants with increasing antibody titer > 4 times and/or percentage of infants with transition of seronegative to seropositive
Seroconversion | 28 days after immunization
  Comparison of GMT, seroprotection, percentage of subjects with increasing antibody titer > 4 times and/ or percentage of subjects with transition of seronegative to seropositive following primary series of investigational product compare to control.

CONTACTS AND LOCATIONS:
Overall Officials: Eddy Fadliyana, Principal Investigator — Hasan Sadikin General Hospital
Locations (3):
- Indonesia (3):
  - Garuda Primary Health Centre, Bandung, West Java
  - Ibrahim Adjie Primary Health Centre, Bandung, West Java
  - Puter Primary Health Care, Bandung, West Java